CLINICAL TRIAL: NCT01886859
Title: A Dose Escalation Study of Ibrutinib With Lenalidomide for Relapsed and Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Lenalidomide and Ibrutinib in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00888; NCI-2013-00888 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-0110; 12-164; 9254 (Other: University of Colorado Hospital); 9254 (Other: CTEP); P30CA046934 (NIH); P50CA140158 (NIH); U01CA076576 (NIH); UM1CA186688 (NIH); UM1CA186712 (NIH)
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Recurrent B-Cell Prolymphocytic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory B-Cell Prolymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Prolymphocytic, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; Lenalidomide

ARMS (1):
- Treatment (ibrutinib and lenalidomide) (Experimental): Patients receive a run-up cycle of ibrutinib PO daily on days 1-28. Patients then receive ibrutinib PO and lenalidomide PO daily on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. After 12 cycles, patients who have achieved CR/CRi, nodular PR, partial remission with persistent lymphocytosis, partial remission, or who have stable disease discontinue lenalidomide and continue ibrutinib.
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase I trial studies the side effects and best dose of lenalidomide when given together with ibrutinib in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma that has returned after a period of improvement (relapsed) or does not respond to treatment (refractory). Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving lenalidomide together with ibrutinib may work better in treating chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the safety, tolerability and maximum tolerated dose (MTD) of lenalidomide when used in combination with ibrutinib in adults with relapsed or refractory chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL).

SECONDARY OBJECTIVES:

I. To determine the response rate and response duration in relapsed and refractory CLL/SLL patients with ibrutinib and lenalidomide.

II. To characterize the plasma pharmacokinetic (PK) interaction between ibrutinib and lenalidomide.

III. To explore whether pharmacogenetic studies can predict response, resistance or toxicity to ibrutinib and lenalidomide.

IV. To explore the ability of ibrutinib to occupy its targets (Bruton's tyrosine kinase [BTK] in B-cells and interleukin-2 inducible kinase [ITK] in T-cells), and whether co-administration with lenalidomide influences this binding.

V. To explore the early and late immunologic consequences of combining ibrutinib with lenalidomide in relapsed and refractory CLL.

VI. To explore the impact of ibrutinib and lenalidomide on ras homolog family member H (RhoH) expression and whether baseline RhoH expression predicts outcomes with this regimen.

VII. To explore mechanisms of resistance to ibrutinib. VIII. To explore the influence of traditional and new CLL/SLL clinical and laboratory prognostic factors on response to ibrutinib and lenalidomide.

OUTLINE: This is a dose-escalation study of lenalidomide.

Patients receive a run-up cycle of ibrutinib orally (PO) daily on days 1-28. Patients then receive ibrutinib PO and lenalidomide PO daily on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. After 12 cycles, patients who have achieved complete remission (CR)/CR with incomplete marrow recovery (CRi), nodular partial remission (PR), partial remission with persistent lymphocytosis, partial remission, or who have stable disease discontinue lenalidomide and continue ibrutinib.

After completion of study treatment, patients are followed up for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of CLL/SLL or B-cell prolymphocytic leukemia, as defined by the World Health Organization (WHO)
* During dose escalation, patients must have received at least one prior therapy, need additional cytoreduction, and meet criteria for relapsed or refractory disease; relapsed disease is defined as a patient who previously achieved a CR or a PR, but after a period of six or more months demonstrates evidence of disease progression; refractory disease is defined as progression within six months of the last anti-leukemic therapy, or any response less than a CR or PR; patients who are previously untreated, and do not wish to receive chemotherapy or immunotherapy, are eligible for the dose expansion portion of the study
* Patients may have not received treatment for 28 days before the first day of the study protocol (dose escalation only)
* Estimated life expectancy greater than two months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Ability to understand and willingness to sign a written informed consent document
* Patients must have acceptable organ and marrow function, which should be present independent of growth factor or transfusion support for at least 7 days prior to first dose of study drug, with the exception of pegylated G-CSF (pegfilgrastim) and darbopoeitin which require a 14-day period between dosing and first dose of study drug
* Absolute neutrophil count (ANC) >= 750 cells/uL (0.75 x 10^9/L)
* Platelets >= 50,000 cells/uL (50 x 10^9/L)
* Hemoglobin > 8 mg/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless Gilbert's syndrome or disease infiltration of the liver is present
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x ULN
* Creatinine < 2.0 x ULN or creatinine clearance (estimated [est.] glomerular filtration rate [GFR] [Cockcroft-Gault]) >= 30 mL/min
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time (PTT)/activated partial thromboplastin time (aPTT) < 1.5 x ULN
* The effects of ibrutinib on the developing human fetus are unknown; lenalidomide is likely to be teratogenic; therefore, females of childbearing potential (FCBP) must have a negative pregnancy test (sensitivity of at least 25 mIU/mL) performed once before ibrutinib and a total of two negative tests before initiating lenalidomide; a FCBP is a female who: 1) has achieved menarche at some point; 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); the pre-ibrutinib pregnancy test will be initiated at enrollment; the first pre- lenalidomide test will be performed within 10-14 days of starting lenalidomide (cycle 0, day 15), and the second pre-lenalidomide test (3rd total test) will be within 24 hours of the first dose of lenalidomide; the patient may not receive lenalidomide until the study doctor has verified that the results of these pregnancy tests are negative; pregnancy tests (if applicable) are then to be conducted weekly during the first month, and monthly thereafter in women with a regular menstrual cycle, as well as at study discontinuation, and at day 28 following study discontinuation; if menstrual cycles are irregular, pregnancy testing will be conducted weekly for the first month, and then every 14 days while on the study, at study discontinuation, and at days 14 and 28 following study drug discontinuation; pregnancy testing and counseling are to be performed if a patient misses her period or if there is any abnormality in menstrual bleeding; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately; further, FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; male and female patients must agree to use highly effective methods of birth control (e.g. condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete sexual abstinence, or sterilized partner) during the period of therapy and for 90 days after the last dose of study drug; all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure

Exclusion Criteria:

* Prior therapy with Bruton's tyrosine kinase (BTK) inhibitor
* Concurrent treatment with other investigational or anti-neoplastic agents
* Patients requiring daily corticosteroids at a prednisone equivalent of > 20 mg daily should not be enrolled; if corticosteroids can be discontinued (or reduced to < 20 mg per day of prednisone or equivalent), the discontinuation or dose reduction should be done at least 7 days prior to first dose
* Chemotherapy =< 21 days prior to first administration of study treatment and/or monoclonal antibody =< 6 weeks prior to first administration of study treatment; immunotherapy, radiotherapy or experimental therapy within 28 days of first day of study drug dosing, or within six weeks of first day of study drug dosing in the event that nitrosoureas or mitomycin were used; concurrent systemic immunosuppressant therapy other than corticosteroids (e.g. cyclosporine A, tacrolimus, etc) must be discontinued within 28 days of the first dose of study drug
* Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, or any class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification, or history of myocardial infarction, unstable angina or acute coronary syndrome within 6 months prior to on-study registration
* Uncontrolled psychiatric illness that would limit compliance with study requirements
* Central nervous system disease involvement; these patients should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of prior malignancy, with the exception of the following:

  * Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to screening, and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanomatous skin cancer or lentigo maligna melanoma without current evidence of disease
  * Adequately treated cervical carcinoma in situ without current evidence of disease
* Serologic status reflecting active hepatitis B or C infection; patients that are hepatitis B core antibody, hepatitis B surface antigen (HBsAg) or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment; PCR positive patients will be excluded
* Active infection at initiation of study; recent infections requiring systemic treatment need to have completed therapy > 14 days before the first dose of study drug
* Major surgery within 4 weeks or minor surgery within 7 days of the first day of study drug dosing
* Unable to swallow capsules or disease significantly affecting gastrointestinal function or resection of the stomach or small bowel, or symptomatic inflammatory bowel disease or ulcerative colitis or partial or complete bowel obstruction
* Prior allogeneic stem cell transplantation
* Active, uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura (ITP)
* Presence of transfusion-dependent thrombocytopenia or a history of bleeding disorders or clinical conditions (e.g. gastrointestinal [GI] bleeding or constitutional disorders) that may increase risk of life-threatening bleeding when thrombocytopenic
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib or lenalidomide
* Patients who received a strong cytochrome P450 (CYP) 3A inhibitor within 7 days prior to the first dose of ibrutinib or patients who require continuous treatment with a strong CYP3A inhibitor
* Requires or is receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g.: phenprocoumon) within 28 days of the first dose of study drug
* Pregnant women are excluded from this study because ibrutinib and lenalidomide have the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ibrutinib and lenalidomide, breastfeeding should be discontinued if the mother is treated with either agent, and for 30 days after discontinuation of therapy
* Current life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, or put the study at risk
* Human immunodeficiency virus (HIV)-positive patients with cluster of differentiation 4 (CD4) counts less than the lower limit of institutional normal
* HIV-positive patients requiring antivirals which are cytochrome P450 (CYP) interactive with the investigational agents (CYP3A4 strong inducers and inhibitors)
* Other laboratory abnormalities that, in the opinion of the investigator, would compromise the patient's safety or interfere with data interpretation
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 5), grade =< 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* Unwilling or unable to participate in all required study evaluations and procedures
* Currently active, clinically significant hepatic impairment (>= moderate hepatic impairment according to the National Cancer Institute (NCI)/Child Pugh classification)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-04-26 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of lenalidomide when combined with ibrutinib | 28 days
  Defined as the highest dose in which less than or equal to 1/6 patients have dose limiting toxicity. Assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. All patient safety information collected will be summarized using descriptive statistics (number of non-missing values, mean, median, standard deviation, minimum and maximum) for continuous variables and counts and percentages for categorical variables, where applicable.

SECONDARY OUTCOMES:
Response rates | Up to 12 months
  Response rates will be calculated based on all the intention-to-treat subjects and reported along with its exact 95% confidence interval.
Remission/response duration | Up to 90 days
  Remission/response duration is measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Response duration will be calculated, and the mean, median, minimum, and maximum values will be reported.

OTHER OUTCOMES:
Non-compartmental areas under the curve (AUCs) for ibrutinib | Up to day 1 of cycle 2
  The impact of lenalidomide on pharmacokinetics of ibrutinib will be evaluated by comparisons of non-compartmental AUCs for ibrutinib on cycle 0, day 8 versus cycle 2, day 1.
Ability of ibrutinib to bind to its targets | Up to day 1 of cycle 2
  The impact of lenalidomide on ibrutinib binding to Bruton's tyrosine kinase and interleukin-2 inducible kinase will be evaluated, and the mechanistic interactions between the two agents will be investigated.
Percentage of occupancy | Up to day 1 of cycle 2
  Defined as the ratio between the signal pre-dose and the signal post-dose. More than 95% occupancy is defined as full occupancy.
Change in Rho guanosine triphosphate (GTP)ase levels | Baseline to up to day 1 of cycle 2
  Comparison of Rho GTPase expression and activation levels, as well as migration before and after treatment with lenalidomide, will be performed using a paired Student t test. The predictive power of the clinical and laboratory values measured for purposes of biomarker discover will be assessed by a multiple comparison analysis of variance test.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Pollyea, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of Colorado Hospital, Aurora, Colorado
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio